CLINICAL TRIAL: NCT02217072
Title: A Randomized Controlled Trial of Educational Support Interventions for Children in Care
Brief Title: Educational Support Interventions for Children in Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VIVE - The Danish Center for Social Science Research (Other)
Collaborators: Ministry of Social Affairs (Ambiguous)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFI 2691
Record Dates: First submitted 2014-07-28; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Learning Problems
Keywords: academic performance; cognitive development; children in care; prevention of school failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Control
- Parents as Tutors (Experimental): Educational support intervention
  Interventions: Behavioral: Parents as Tutors
- school intervention (Experimental): Educational support intervention
  Interventions: Behavioral: School intervention

INTERVENTIONS:
Behavioral: School intervention — A school-based intervention that builds on the promising Swedish programme SkolFam, but is adapted to a Danish school context. The two main components of the programme are a) comprehensive assessment of the child, involving testing of the child's cognitive and academic abilities and difficulties as well as an evaluation of the child's behaviour, school-related social relations and well-being, and b) a systematic and individually targeted intervention plan, made in collaboration between a psychologist, the teachers, and a special educational teacher at the school (e.g., the reading counsellor).
  Arms: school intervention
Behavioral: Parents as Tutors — A home-based intervention, comprising a structured tutoring programme that allows foster parents to systematically support the foster child's school performance. Foster parents will attend an introductory tutor training seminar at which they will be introduced to relevant theory on learning and counselled on tutoring practice. The intervention itself is designed to provide approximately three hours per week of individual home-based tutoring for a period of 40 weeks.
  Arms: Parents as Tutors

SUMMARY:
A Randomized controlled study of two different educational support interventions developed for children in foster care (age 6-13).

DETAILED DESCRIPTION:
A Randomized controlled study of two different educational support interventions developed for children in foster care (age 6-13). One intervention is school-based and involves a team of professionals at the child's school, and the other is a home-based tutoring intervention provided by the foster parents. The participants in the study are assigned to three groups (the two intervention groups and control group). Based on power calculation we aim to recruit approximately 180-200 foster children, their foster parents and public schools to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* age 6-13
* fostercare placement
* placement in a participating municipality

Exclusion Criteria:

* persuasive developmental disorders
* special education students

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 190 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Academic performance | 17 months after intervention start
  Reading test and mathematical test

SECONDARY OUTCOMES:
Cognitive functions | 17 months after intervention start
  Wechsler Intelligence Scale for Children IV and Contingency Naming Test

OTHER OUTCOMES:
well-being | 17 months after intervention start
  The Strengths and Difficulties Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Misja Eiberg, Ph.d. fellow, Principal Investigator — SFI - The Danish National Centre for Social Research
Locations (1):
- SFI - The Danish National Centre for Social Research, Copenhagen, Denmark